CLINICAL TRIAL: NCT02319759
Title: A Phase 2a, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Guselkumab in the Treatment of Subjects With Active Psoriatic Arthritis
Brief Title: Efficacy and Safety Study of Guselkumab in the Treatment of Participants With Active Psoriatic Arthritis (PsA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR105964; 2014-003697-17 (EudraCT Number); CNTO1959PSA2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Guselkumab; Ustekinumab; Placebo
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Guselkumab (Experimental): Participants will receive guselkumab 100 milligram (mg) subcutaneous injection (injected under the skin by way of a needle) at Weeks 0, 4, 12, 20, 28, 36, and 44, and placebo for guselkumab at Week 24 to maintain the blind. Participants who enter early escape at Week 16 will switch to open label therapy with ustekinumab 45 mg or 90 mg at Weeks 16, 20, 32, and 44 based on the approved dosage in the particular country of the study.
  Interventions: Drug: Guselkumab; Drug: Ustekinumab; Drug: Placebo
- Placebo (Experimental): Participants will receive placebo for guselkumab at Weeks 0, 4, 12, and 20, and guselkumab 100 mg subcutaneous injection at Weeks 24, 28, 36, and 44. Participants who enter early escape at Week 16 will switch to open label therapy with ustekinumab 45 mg or 90 mg at Weeks 16, 20, 32, and 44 based on the approved dosage in the particular country of the study.
  Interventions: Drug: Guselkumab; Drug: Ustekinumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — In the guselkumab group, Guselkumab 100 mg subcutaneous injection will be administered at Weeks 0, 4, 12, 20, 28, 36 and 44. In the placebo group, guselkumab 100 mg subcutaneous injection will be administered at Weeks 24, 28, 36 and 44 for participants remaining on placebo at Week 24.
Drug: Ustekinumab — In both placebo and guselkumab groups, if the participants qualify for early escape, they will switch to receive ustekinumab 45 mg or 90 mg subcutaneous injection at Weeks 16, 20, 32, and 44 based on the approved dosage in the particular country of the study.
Drug: Placebo — In placebo group, Placebo subcutaneous injection will be administered at Weeks 0, 4, 12, and 20. In guselkumab group, placebo subcutaneous injection will be administered at Week 24 to maintain the blind.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of guselkumab in participants with Active Psoriatic Arthritis (PsA).

DETAILED DESCRIPTION:
This is a multi-center (more than one clinical site will work on a medical research study), randomized (study medication assigned to participants by chance), double-blind (neither investigator nor participant knows which treatment the participant receives), placebo-controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial) study to determine the efficacy and safety of guselkumab in participants with PsA. The study will consist of 4 parts: Screening period (6 weeks), a double-blind treatment period (consists of guselkumab and placebo treatment for 24 weeks), an active treatment period (guselkumab for 20 weeks), and follow-up period (12 weeks). The maximal study duration for a participant will not exceed 62 weeks including the Screening period. Eligible participants will be randomly assigned to one of two groups in a 2:1 ratio to either receive Guselkumab 100 milligram (mg) at Weeks 0, 4 then every 8 weeks or Placebo at Weeks 0, 4 then every 8 weeks until Week 24. At week 24, participants remaining in the placebo group will start to receive guselkumab 100 mg at Weeks 24, 28, 36 and 44. Participants in both treatment groups who have less than (<) 5 percent (%) improvement from baseline in both tender and swollen joint counts at Week 16 will qualify for early escape and will switch to open-label therapy with ustekinumab 45 mg or 90 mg at Weeks 16, 20, 32, and 44 based on the approved dosage for the PsA indication in the particular country of study. The efficacy will be assessed primarily by measuring percentage of participants who achieve an American College of Rheumatology (ACR) 20 Response at Week 24. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Has had Psoriatic Arthritis (PsA) for at least 6 months before the first administration of study drug and meet classification criteria for Psoriatic Arthritis (CASPAR) at Screening
* Had active PsA as defined by:

  1. At least 3 swollen joints and at least 3 tender joints at Screening and at baseline
  2. C-reactive protein (CRP) greater than or equal to (>=) 0.3 milligram (mg)/deciliter (dL) at Screening from the central laboratory
* Has at least 1 of the PsA subsets: distal interphalangeal joint involvement, polyarticular arthritis with absence of rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis
* Has plaque psoriasis with body surface area (BSA) involvement greater than or equal to (>=) 3% at Screening and baseline
* Has active PsA despite current or previous non-biologic disease-modifying antirheumatic drugs (DMARD), oral corticosteroid, and/or nonsteroidal anti-inflammatory drug (NSAID) therapy
* If using methotrexate (MTX), oral corticosteroids or NSAIDs, the dose must be stable

Exclusion Criteria:

* Have other inflammatory diseases that might confound the evaluations of benefit of guselkumab therapy, including but not limited to rheumatoid arthritis (RA), ankylosing spondylitis (AS), systemic lupus erythematosus, or Lyme disease
* Has previously received guselkumab or ustekinumab
* Has received more than 1 type of biologic anti-tumor necrosis factor (TNF) agent previously
* Have received infliximab (or its biosimilars) or golimumab intraveneous (IV) within 12 weeks before the first administration of study drug
* Have received adalimumab (or its biosimilars), golimumab subcutaneous (SC), certolizumab pegol or etanercept (or its biosimilars) within 8 weeks before the first administration of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2017-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (41):
- United States (12):
  - Huntsville, Alabama
  - Trumbull, Connecticut
  - Clearwater, Florida
  - Tampa, Florida
  - Sandy Springs, Georgia
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Edina, Minnesota
  - St Louis, Missouri
  - Wyomissing, Pennsylvania
  - Jackson, Tennessee
  - Arlington, Virginia
- Canada (4):
  - Barrie, Ontario
  - London, Ontario
  - Peterborough, Ontario
  - Waterloo, Ontario
- Germany (6):
  - Berlin
  - Cologne
  - Hamburg
  - Herne
  - Kiel
  - Lübeck
- Poland (4):
  - Bialystok
  - Elblag
  - Poznan
  - Warsaw
- Bucharest, Romania
- Russia (9):
  - Bataysk
  - Moscow
  - Novosibirsk
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Ufa
  - Ulyanovsk
  - Yaroslavl
- Spain (5):
  - Barcelona
  - Madrid
  - Sabadell
  - Santiago de Compostela
  - Seville

REFERENCES:
- [Derived] Strober B, Coates LC, Lebwohl MG, Deodhar A, Leibowitz E, Rowland K, Kollmeier AP, Miller M, Wang Y, Li S, Chakravarty SD, Chan D, Shawi M, Yang YW, Thaҫi D, Rahman P. Long-Term Safety of Guselkumab in Patients with Psoriatic Disease: An Integrated Analysis of Eleven Phase II/III Clinical Studies in Psoriasis and Psoriatic Arthritis. Drug Saf. 2024 Jan;47(1):39-57. doi: 10.1007/s40264-023-01361-w. Epub 2023 Oct 31. PMID 37906417
- [Derived] Rahman P, Boehncke WH, Mease PJ, Gottlieb AB, McInnes IB, Shawi M, Wang Y, Sheng S, Kollmeier AP, Theander E, Yu J, Leibowitz E, Marrache AM, Coates LC. Safety of Guselkumab With and Without Prior Tumor Necrosis Factor Inhibitor Treatment: Pooled Results Across 4 Studies in Patients With Psoriatic Arthritis. J Rheumatol. 2023 Jun;50(6):769-780. doi: 10.3899/jrheum.220928. Epub 2023 Jan 15. PMID 36642439
- [Derived] Mease PJ, Gladman DD, Deodhar A, McGonagle DG, Nash P, Boehncke WH, Gottlieb A, Xu XL, Xu S, Hsia EC, Karyekar CS, Helliwell PS. Impact of guselkumab, an interleukin-23 p19 subunit inhibitor, on enthesitis and dactylitis in patients with moderate to severe psoriatic arthritis: results from a randomised, placebo-controlled, phase II study. RMD Open. 2020 Jul;6(2):e001217. doi: 10.1136/rmdopen-2020-001217. PMID 32665433
- [Derived] Helliwell PS, Deodhar A, Gottlieb AB, Boehncke WH, Xu XL, Xu S, Wang Y, Hsia EC, Gladman DD, Ritchlin CT. Composite Measures of Disease Activity in Psoriatic Arthritis: Comparative Instrument Performance Based on the Efficacy of Guselkumab in an Interventional Phase II Trial. Arthritis Care Res (Hoboken). 2020 Nov;72(11):1579-1588. doi: 10.1002/acr.24046. PMID 31421033
- [Derived] Deodhar A, Gottlieb AB, Boehncke WH, Dong B, Wang Y, Zhuang Y, Barchuk W, Xu XL, Hsia EC; CNTO1959PSA2001 Study Group. Efficacy and safety of guselkumab in patients with active psoriatic arthritis: a randomised, double-blind, placebo-controlled, phase 2 study. Lancet. 2018 Jun 2;391(10136):2213-2224. doi: 10.1016/S0140-6736(18)30952-8. Epub 2018 Jun 1. PMID 29893222

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Week 0 to Week 24): Participants were randomized at Week 0 to receive placebo matched to guselkumab subcutaneous injections at Weeks 0, 4, 12 and 20.
- Placebo to Guselkumab (Week 24 to Week 56): Participants who received placebo matched to guselkumab subcutaneous injections at Weeks 0, 4, 12 and 20 received guselkumab 100 milligram (mg) subcutaneous injections at Weeks 24, 28, 36 and 44, with a final follow-up at Week 56.
- Guselkumab (Week 0 to Week 56): Participants were randomized to receive guselkumab 100 mg subcutaneous injections at Weeks 0, 4, 12, 20, 28, 36 and 44, and placebo at Week 24, with a final follow-up at Week 56.
- Placebo to Ustekinumab (Week 16 to Week 56): Participants who were randomized to receive placebo matched to guselkumab subcutaneous injections at Weeks 0, 4 and 12, and had less than (<) 5 percent (%) improvement from baseline in both tender and swollen joint counts at Week 16 were qualified for early escape (EE) and switched to open-label ustekinumab subcutaneous injections at the approved dosage (45 mg or 90 mg) for psoriatic arthritis (PsA) in the particular country of the study at Weeks 16, 20, 32 and 44, with a final follow-up at Week 56.
- Guselkumab to Ustekinumab (Week 16 to Week 56): Participants who were randomized to receive guselkumab 100 mg subcutaneous injections at Weeks 0, 4, 12 and had <5% improvement from baseline in both tender and swollen joint counts at Week 16 were qualified for EE and switched to open-label ustekinumab subcutaneous injections at the approved dosage (45 mg or 90 mg) for PsA in the particular country of the study at Weeks 16, 20, 32 and 44, with a final follow-up at Week 56.
Period: Week 0 - 16
Arm/Group | Placebo (Week 0 to Week 24) | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 0 to Week 56) | Placebo to Ustekinumab (Week 16 to Week 56) | Guselkumab to Ustekinumab (Week 16 to Week 56)
Started | 49 | 0 | 100 | 0 | 0
Completed | 48 | 0 | 99 | 0 | 0
Not Completed | 1 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — Not met all Inclusion Criteria | 0 | 0 | 1 | 0 | 0
Period: Week 16 - 24
Arm/Group | Placebo (Week 0 to Week 24) | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 0 to Week 56) | Placebo to Ustekinumab (Week 16 to Week 56) | Guselkumab to Ustekinumab (Week 16 to Week 56)
Started | 31 | 0 | 89 | 17 | 10
Completed | 29 | 0 | 86 | 17 | 10
Not Completed | 2 | 0 | 3 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0
Period: Week 24 - 56
Arm/Group | Placebo (Week 0 to Week 24) | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 0 to Week 56) | Placebo to Ustekinumab (Week 16 to Week 56) | Guselkumab to Ustekinumab (Week 16 to Week 56)
Started | 0 | 29 | 86 | 17 | 10
Completed | 0 | 28 | 84 | 15 | 8
Not Completed | 0 | 1 | 2 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants were randomized to receive placebo matched to guselkumab subcutaneous injections at Weeks 0, 4, 12 and 20 and guselkumab 100 milligram (mg) subcutaneous injection at Weeks 24, 28, 36 and 44.
- Guselkumab: Participants were randomized to receive guselkumab 100 mg subcutaneous injections at Weeks 0, 4, 12, 20, 28, 36 and 44, and placebo at Week 24, with a final follow-up at Week 56.
- Total: Total of all reporting groups
Arm/Group | Placebo | Guselkumab | Total
Number analyzed (Participants) | 49 | 100 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (12.43) | 47.4 (12.83) | 46.3 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 48 | 73
  Male | 24 | 52 | 76
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 2 | 4 | 6
  Germany | 2 | 2 | 4
  Spain | 3 | 6 | 9
  Poland | 12 | 13 | 25
  Romania | 1 | 4 | 5
  Russia | 25 | 64 | 89
  United States | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) 20 Response at Week 24
Description: ACR 20 response: at least 20% improvement from baseline in both swollen joint (66 joints) and tender joint (68 joints) counts and at least 20% improvement from baseline in 3 of following 5 assessments: patient's assessment of pain (VAS: 0-100 millimeter [mm], 0=no pain and 100=worst possible pain), patient's global assessment of disease activity on arthritis (VAS:0-100mm, 0=excellent and 100=poor), physician's global assessment of disease activity (VAS:0-100mm; 0=no arthritis activity and 100 = extremely active arthritis), patient's assessment of physical function measured by HAQ-DI (defined as a 20-question instrument assessing 8 functional areas;derived HAQ-DI ranges from 0=no difficulty, to 3=inability to perform a task in that area) and serum CRP. Treatment Failure (TF) criteria: Discontinued study drug due to lack of efficacy or worsening of PsA, initiated or increased dose of methotrexate or oral corticosteroids, or initiated prohibited PsA treatments. FAS is full analysis set.
Time Frame: Week 24
Population: FAS (up to Week 24): participants randomized and received 1 dose of study drug per assigned treatment regardless of actual treatments received. Data after meeting TF criteria or after EE to ustekinumab and missing data are imputed as non-responders. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants were randomized at Week 0 to receive placebo matched to guselkumab subcutaneous injections at Weeks 0, 4, 12 and 20.
- Guselkumab: Participants were randomized at Week 0 to receive guselkumab 100 mg subcutaneous injections at Weeks 0, 4, 12 and 20.
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
percentage of participants | 18.4 | 58.0
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Percent difference = 39.7, 95% CI 2-sided [25.3 to 54.1]

2. Secondary Outcome: Percentage of Participants Who Achieved a Psoriasis Area and Severity Index (PASI)-75 Response at Week 24
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72 (worst condition). PASI 75 response was defined as at least a 75% reduction in PASI relative to Baseline. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Time Frame: Week 24
Population: Full Analysis Set (FAS) (up to Week 24). Data after EE to ustekinumab and missing data were imputed using last observation carried forward (LOCF). Here 'N' (number of participants analyzed) included all participants who were evaluable for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 48 | 98
percentage of participants | 12.5 | 78.6
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Percentage (%) Difference = 66.1, 95% CI 2-sided [53.8 to 78.4]

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24
Description: Change from baseline in HAQ-DI score is a measure of the change in the physical function, where a negative change reflects an improvement and a positive change reflects worsening of physical function. HAQ-DI is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0 indicating no difficulty, to 3 indicating inability to perform a task in that area (that is, lower scores are indicative of better functioning). The total HAQ-DI score ranges from 0-24 with lower score indicating better functioning.
Time Frame: Baseline and Week 24
Population: FAS (up to Week 24). Data after EE to ustekinumab and missing data were imputed using LOCF. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
units on a scale | -0.06 (0.530) | -0.42 (0.512)
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; Test type: Superiority; p < 0.001, MMRM; MMRM stands for Mixed-effects Model Repeated Measures; Least Square Mean Difference = -0.31, 95% CI 2-sided [-0.471 to -0.148]

4. Secondary Outcome: Percentage of Participants Who Achieved an ACR 20 Response at Week 16
Description: ACR 20 response is defined as at least 20 percent (%) improvement from baseline in both swollen joint (66 joints) and tender joint (68 joints) counts and at least 20% improvement from baseline in 3 of following 5 assessments: patient's assessment of pain (visual analog scale [VAS]: 0-100 millimeter [mm]; 0=no pain and 100=worst possible pain), patient's global assessment of disease activity on arthritis (VAS: 0-100 mm, 0=excellent and 100=poor), physician's global assessment of disease activity (VAS: 0-100mm; 0=no arthritis activity and 100 = extremely active arthritis), patient's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas;derived HAQ-DI ranges from 0 indicating no difficulty, to 3 indicating inability to perform a task in that area) and serum C-Reactive Protein (CRP).
Time Frame: Week 16
Population: FAS (up to Week 24). Data after meeting TF criteria or after EE to ustekinumab and missing data are imputed as non-responders. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
percentage of participants | 16.3 | 60.0

5. Secondary Outcome: Percentage of Participants Who an Achieved ACR 50 Response at Week 24
Description: ACR 50 response is defined as at least 50 % improvement from baseline in both swollen joint (66 joints) and tender joint (68 joints) counts and at least 50% improvement from baseline in 3 of following 5 assessments: patient's assessment of pain (VAS:0-100 mm; 0=no pain and 100=worst possible pain), patient's global assessment of disease activity on arthritis (VAS:0-100mm; 0=excellent and 100=poor), physician's global assessment of disease activity (VAS: 0-100mm; 0=no arthritis activity and 100 = extremely active arthritis), patient's assessment of physical function measured by HAQ-DI (defined as a 20-question instrument assessing 8 functional areas;derived HAQ-DI ranges from 0 indicating no difficulty, to 3 indicating inability to perform a task in that area) and serum CRP.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
percentage of participants | 10.2 | 34.0

6. Secondary Outcome: Percent Change From Baseline in Leeds Enthesitis Index (LEI) Scores Among Participants With Enthesitis at Week 24
Description: Enthesitis was assessed using the Leeds Enthesitis Index (LEI). The LEI was developed to assess enthesitis in participants with psoriatic arthritis (PsA), and evaluates the presence (score of 1) or absence of pain (score of 0) by applying local pressure to Lateral elbow epicondyle, left and right, Medial femoral condyle, left and right, and Achilles tendon insertion, left and right. LEI scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness).
Time Frame: Baseline and Week 24
Population: FAS (up to Week 24) and had enthesitis at baseline. Data after EE to ustekinumab or missing data are imputed using LOCF. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 31 | 76
percent change | -33.33 [-100.0 to 0.0] | -100.00 [-100.0 to -10.0]

7. Secondary Outcome: Percent Change From Baseline in Dactylitis Scores Among Participants With Dactylitis at Baseline at Week 24
Description: Dactylitis is characterized by swelling of the entire finger or toe. The severity of dactylitis is scored on a scale of 0-3, where 0, 1, 2, 3 indicates none, mild, moderate, severe, respectively in each digit of the hands and feet. The range of total dactylitis scores for a participant is 0-60. Higher score indicates more severe dactylitis.
Time Frame: Baseline and Week 24
Population: FAS (up to Week 24) and had dactylitis at baseline. Data after EE to ustekinumab or missing data were imputed using LOCF. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 23 | 58
percent change | -33.33 [-66.7 to 0.0] | -100.00 [-100.0 to -50.0]

8. Secondary Outcome: Percentage of Participants Who Achieved ACR 20, ACR 50, and ACR 70 Responses at Weeks 4, 8, 12, 16, 20, and 24
Description: ACR 20, 50, and 70 response is defined as at least 20%, 50%, and 70% improvement from baseline in swollen joint (66 joints) and tender joint (68 joints) counts and at least 20%, 50%, and 70% improvement from baseline in 3 of following 5 assessments: patient's assessment of pain (VAS: 0-100mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity on arthritis (VAS: 0-100mm; 0=excellent and 100=poor), physician's global assessment of disease activity (VAS: 0-100mm; 0=no arthritis activity and 100= extremely active arthritis), patient's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas;derived HAQ-DI ranges from 0 indicating no difficulty, to 3 indicating inability to perform a task in that area) and serum C-Reactive Protein (CRP).
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
percentage of participants
  Week 4: ACR 20 responders | 0 | 21.0
  Week 4: ACR 50 responders | 0 | 1.0
  Week 4: ACR 70 responders | 0 | 0
  Week 8: ACR 20 responders | 22.4 | 42.0
  Week 8: ACR 50 responders | 6.1 | 12.0
  Week 8: ACR 70 responders | 2.0 | 4.0
  Week 12: ACR 20 responders | 12.2 | 49.0
  Week 12: ACR 50 responders | 6.1 | 15.0
  Week 12: ACR 70 responders | 0 | 7.0
  Week 16: ACR 20 responders | 16.3 | 60.0
  Week 16: ACR 50 responders | 6.1 | 30.0
  Week 16: ACR 70 responders | 4.1 | 9.0
  Week 20: ACR 20 responders | 22.4 | 63.0
  Week 20: ACR 50 responders | 10.2 | 37.0
  Week 20: ACR 70 responders | 2.0 | 11.0
  Week 24: ACR 20 responders | 18.4 | 58.0
  Week 24: ACR 50 responders | 10.2 | 34.0
  Week 24: ACR 70 responders | 2.0 | 14.0

9. Secondary Outcome: Percentage of Participants Who Achieved ACR 20, ACR 50, and ACR 70 Responses at Weeks 24, 28, 32, 36, 44, and 56
Description: ACR 20, ACR 50 and ACR 70 response is defined as at least 20%, 50%, and 70% improvement from baseline in swollen joint (66 joints) and tender joint (68 joints) counts and at least 20%, 50%, and 70% improvement from baseline in 3 of following 5 assessments: patient's assessment of pain (VAS: 0-100mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity on arthritis (VAS: 0-100mm; 0=excellent and 100=poor), physician's global assessment of disease activity (VAS; 0-100mm; 0=no arthritis activity and 100 = extremely active arthritis), patient's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas;derived HAQ-DI ranges from 0 indicating no difficulty, to 3 indicating inability to perform a task in that area) and serum C-Reactive Protein (CRP). As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Time Frame: Weeks 24, 28, 32, 36, 44, and 56
Population: Post Week 24 Efficacy analysis set: included all randomized participants who did not EE to ustekinumab at Week 24, with observed data. Here 'n' (number analyzed) included all participants who were evaluable at specified timepoints.
Measure: Number; unit: percentage of participants
Groups:
- Placebo to Guselkumab (Week 24 to Week 56): Participants who were randomized to receive placebo matched to guselkumab at Weeks 0, 4, 12 and 20 received guselkumab 100 mg subcutaneous injection at Weeks 24, 28, 36 and 44.
- Guselkumab (Week 24 to Week 52): Participants were randomized to receive guselkumab 100 mg subcutaneous injections at Weeks 0, 4, 12, 20, 28, 36 and 44, and matched placebo at Week 24.
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
percentage of participants
  Week 24: ACR 20 responders | 31.0 | 66.3
  Week 24: ACR 50 responders | 17.2 | 39.5
  Week 24: ACR 70 responders | 3.4 | 16.3
  Week 28: ACR 20 responders: number analyzed (Participants) | 28 | 85
  Week 28: ACR 20 responders | 57.1 | 75.3
  Week 28: ACR 50 responders: number analyzed (Participants) | 28 | 85
  Week 28: ACR 50 responders | 28.6 | 44.7
  Week 28: ACR 70 responders: number analyzed (Participants) | 28 | 85
  Week 28: ACR 70 responders | 14.3 | 30.6
  Week 32: ACR 20 responders: number analyzed (Participants) | 28 | 84
  Week 32: ACR 20 responders | 60.7 | 75.0
  Week 32: ACR 50 responders: number analyzed (Participants) | 28 | 84
  Week 32: ACR 50 responders | 42.9 | 51.2
  Week 32: ACR 70 responders: number analyzed (Participants) | 28 | 84
  Week 32: ACR 70 responders | 21.4 | 29.8
  Week 36: ACR 20 responders: number analyzed (Participants) | 28 | 84
  Week 36: ACR 20 responders | 71.4 | 73.8
  Week 36: ACR 50 responders: number analyzed (Participants) | 28 | 84
  Week 36: ACR 50 responders | 46.4 | 48.8
  Week 36: ACR 70 responders: number analyzed (Participants) | 27 | 84
  Week 36: ACR 70 responders | 29.6 | 31.0
  Week 44: ACR 20 responders: number analyzed (Participants) | 28 | 84
  Week 44: ACR 20 responders | 75.0 | 77.4
  Week 44: ACR 50 responders: number analyzed (Participants) | 28 | 84
  Week 44: ACR 50 responders | 46.4 | 46.4
  Week 44: ACR 70 responders: number analyzed (Participants) | 28 | 84
  Week 44: ACR 70 responders | 25.0 | 26.2
  Week 56: ACR 20 responders: number analyzed (Participants) | 27 | 83
  Week 56: ACR 20 responders | 81.5 | 73.5
  Week 56: ACR 50 responders: number analyzed (Participants) | 27 | 83
  Week 56: ACR 50 responders | 66.7 | 53.0
  Week 56: ACR 70 responders: number analyzed (Participants) | 28 | 83
  Week 56: ACR 70 responders | 28.6 | 32.5

10. Secondary Outcome: Percent Change From Baseline in the ACR Components at Weeks 12 and 24
Description: The 7 components of ACR response are: swollen joint counts (0-66), tender joint counts (0-68), patient's assessment of pain (PAIN) (VAS:0-100mm; 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (GDPT) on arthritis (VAS:0-100mm; 0=excellent and 100= poor), physician's global assessment of disease activity (GDEV) (VAS: 0-100mm; 0=no arthritis activity and 100 = extremely active arthritis), patient's assessment of physical function measured by HAQ-DI (20-question instrument assessing 8 functional areas (total score of 0-24 with lower score indicating better functioning);derived HAQ-DI ranges from 0 indicating no difficulty, to 3 indicating inability to perform a task in that area) and serum CRP.
Time Frame: Baseline and Weeks 12, 24
Population: FAS (up to Week 24). Data after EE to ustekinumab and missing data were imputed using LOCF. Here 'n' (number analyzed) included all participants who were evaluable at specified timepoints. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
percent change
  Week 12: Swollen joints (0-66) | -29.41 [-50.0 to 0.0] | -64.50 [-93.8 to -30.0]
  Week 12: Tender joints (0-68) | -13.33 [-46.7 to 15.4] | -45.80 [-78.0 to -25.0]
  Week 12: PAIN (VAS, 0-100 mm): number analyzed (Participants) | 49 | 98
  Week 12: PAIN (VAS, 0-100 mm) | 1.79 [-20.0 to 15.6] | -22.05 [-46.1 to -2.6]
  Week 12: GDPT (VAS, 0-100 mm, arthritis) | -11.39 [-41.0 to 9.2] | -55.24 [-74.5 to -22.1]
  Week 12: GDEV (VAS, 0-100 mm) | -11.39 [-41.0 to 9.2] | -55.24 [-74.5 to -22.1]
  Week 12: HAQ-DI score (0-3): number analyzed (Participants) | 47 | 97
  Week 12: HAQ-DI score (0-3) | 0.00 [-25.0 to 8.3] | -21.43 [-40.0 to -6.7]
  Week 12: CRP | -3.95 [-41.3 to 51.2] | -42.95 [-69.8 to 10.7]
  Week 24: Swollen joints (0-66) | -11.76 [-59.1 to 11.8] | -84.11 [-100.0 to -43.2]
  Week 24: Tender joints (0-68) | -5.56 [-53.1 to 30.8] | -51.05 [-89.6 to -23.7]
  Week 24: PAIN (VAS, 0-100 mm): number analyzed (Participants) | 49 | 98
  Week 24: PAIN (VAS, 0-100 mm) | 2.38 [-20.9 to 32.8] | -32.93 [-70.7 to -7.6]
  Week 24: GDPT (VAS, 0-100 mm, arthritis) | -2.22 [-26.8 to 26.1] | -35.53 [-68.2 to -7.2]
  Week 24: GDEV (VAS, 0-100 mm) | -8.86 [-48.1 to 11.1] | -68.47 [-86.6 to -37.0]
  Week 24: HAQ-DI score (0-3): number analyzed (Participants) | 47 | 97
  Week 24: HAQ-DI score (0-3) | -10.00 [-27.3 to 12.5] | -28.57 [-52.9 to -8.3]
  Week 24: CRP | 7.94 [-30.3 to 93.5] | -42.64 [-77.7 to 2.3]

11. Secondary Outcome: Percent Change From Baseline in the ACR Components at Weeks 24, 28, 32, 36, 44 and 56
Description: as for outcome 10
Time Frame: Basline and Weeks 24, 28, 32, 36, 44, 56
Population: Post Week 24 efficacy analysis set, based on observed data. Here 'n' (number analyzed) included all participants who were evaluable at specified timepoints. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
percent change
  Week 24: Swollen joints (0-66) | -33.33 [-80.0 to -11.8] | -85.71 [-100.0 to -63.3]
  Week 28: Swollen joints (0-66): number analyzed (Participants) | 28 | 85
  Week 28: Swollen joints (0-66) | -69.05 [-83.3 to -32.7] | -93.75 [-100.0 to -60.9]
  Week 32: Swollen joints (0-66): number analyzed (Participants) | 28 | 84
  Week 32: Swollen joints (0-66) | -84.91 [-95.8 to -50.0] | -100.00 [-100.0 to -73.9]
  Week 36: Swollen joints (0-66): number analyzed (Participants) | 28 | 84
  Week 36: Swollen joints (0-66) | -79.14 [-100.0 to -57.7] | -93.93 [-100.0 to -66.7]
  Week 44: Swollen joints (0-66): number analyzed (Participants) | 28 | 84
  Week 44: Swollen joints (0-66) | -86.11 [-100.0 to -64.6] | -94.56 [-100.0 to -70.6]
  Week 56: Swollen joints (0-66): number analyzed (Participants) | 27 | 83
  Week 56: Swollen joints (0-66) | -100.00 [-100.0 to -63.6] | -100.00 [-100.0 to -75.0]
  Week 24: Tender joints (0-68) | -50.00 [-74.5 to -14.9] | -72.00 [-90.0 to -45.8]
  Week 28: Tender joints (0-68): number analyzed (Participants) | 28 | 85
  Week 28: Tender joints (0-68) | -65.99 [-83.3 to -17.0] | -74.36 [-91.3 to -50.0]
  Week 32: Tender joints (0-68): number analyzed (Participants) | 28 | 84
  Week 32: Tender joints (0-68) | -71.76 [-86.1 to -27.7] | -79.66 [-92.3 to -50.0]
  Week 36: Tender joints (0-68): number analyzed (Participants) | 28 | 84
  Week 36: Tender joints (0-68) | -81.67 [-91.2 to -27.1] | -73.32 [-94.6 to -50.5]
  Week 44: Tender joints (0-68): number analyzed (Participants) | 28 | 84
  Week 44: Tender joints (0-68) | -86.06 [-93.5 to -50.0] | -77.22 [-97.0 to -49.0]
  Week 56: Tender joints (0-68): number analyzed (Participants) | 27 | 83
  Week 56: Tender joints (0-68) | -80.00 [-93.8 to -51.2] | -77.27 [-100.0 to -58.8]
  Week 24: PAIN (VAS, 0-100 mm): number analyzed (Participants) | 29 | 84
  Week 24: PAIN (VAS, 0-100 mm) | -11.69 [-34.6 to 14.8] | -40.98 [-72.3 to -9.2]
  Week 28: PAIN (VAS, 0-100 mm): number analyzed (Participants) | 28 | 83
  Week 28: PAIN (VAS, 0-100 mm) | -23.52 [-59.7 to 4.4] | -49.40 [-80.9 to -14.1]
  Week 32: PAIN (VAS, 0-100 mm): number analyzed (Participants) | 28 | 82
  Week 32: PAIN (VAS, 0-100 mm) | -51.08 [-70.9 to -4.9] | -50.00 [-78.7 to -22.2]
  Week 36: PAIN (VAS, 0-100 mm): number analyzed (Participants) | 28 | 82
  Week 36: PAIN (VAS, 0-100 mm) | -61.13 [-79.6 to -11.5] | -55.83 [-83.3 to -21.4]
  Week 44: PAIN (VAS, 0-100 mm): number analyzed (Participants) | 28 | 82
  Week 44: PAIN (VAS, 0-100 mm) | -58.76 [-83.9 to -11.4] | -45.50 [-81.0 to -12.5]
  Week 56: PAIN (VAS, 0-100 mm): number analyzed (Participants) | 28 | 81
  Week 56: PAIN (VAS, 0-100 mm) | -71.99 [-85.0 to -31.5] | -52.44 [-85.7 to -13.7]
  Week 24: GDPT (VAS, 0-100 mm, arthritis) | -17.74 [-35.1 to 5.7] | -41.98 [-70.4 to -8.9]
  Week 28: GDPT (VAS, 0-100 mm, arthritis): number analyzed (Participants) | 28 | 85
  Week 28: GDPT (VAS, 0-100 mm, arthritis) | -40.73 [-66.5 to -5.7] | -52.17 [-76.9 to -18.8]
  Week 32: GDPT (VAS, 0-100 mm, arthritis): number analyzed (Participants) | 28 | 84
  Week 32: GDPT (VAS, 0-100 mm, arthritis) | -48.62 [-75.4 to -14.0] | -56.83 [-78.2 to -24.0]
  Week 36: GDPT (VAS, 0-100 mm, arthritis): number analyzed (Participants) | 28 | 84
  Week 36: GDPT (VAS, 0-100 mm, arthritis) | -52.17 [-81.0 to -29.1] | -52.09 [-81.9 to -15.5]
  Week 44: GDPT (VAS, 0-100 mm, arthritis): number analyzed (Participants) | 28 | 84
  Week 44: GDPT (VAS, 0-100 mm, arthritis) | -49.53 [-80.1 to -11.4] | -47.21 [-82.6 to -13.6]
  Week 56: GDPT (VAS, 0-100 mm, arthritis): number analyzed (Participants) | 28 | 83
  Week 56: GDPT (VAS, 0-100 mm, arthritis) | -68.12 [-87.1 to -31.8] | -55.32 [-84.0 to -11.8]
  Week 24: GDEV (VAS, 0-100 mm) | -37.88 [-60.6 to -8.9] | -72.41 [-89.7 to -51.5]
  Week 28: GDEV (VAS, 0-100 mm): number analyzed (Participants) | 27 | 84
  Week 28: GDEV (VAS, 0-100 mm) | -66.07 [-86.6 to -48.6] | -80.26 [-92.2 to -55.9]
  Week 32: GDEV (VAS, 0-100 mm): number analyzed (Participants) | 28 | 83
  Week 32: GDEV (VAS, 0-100 mm) | -71.40 [-88.1 to -56.4] | -82.14 [-93.3 to -60.0]
  Week 36: GDEV (VAS, 0-100 mm): number analyzed (Participants) | 25 | 83
  Week 36: GDEV (VAS, 0-100 mm) | -81.82 [-89.2 to -65.9] | -79.75 [-93.0 to -57.1]
  Week 44: GDEV (VAS, 0-100 mm): number analyzed (Participants) | 28 | 83
  Week 44: GDEV (VAS, 0-100 mm) | -82.41 [-89.8 to -65.0] | -80.00 [-92.1 to -61.2]
  Week 56: GDEV (VAS, 0-100 mm): number analyzed (Participants) | 27 | 81
  Week 56: GDEV (VAS, 0-100 mm) | -86.36 [-94.9 to -74.4] | -83.93 [-93.0 to -54.1]
  Week 24: HAQ-DI score (0-3): number analyzed (Participants) | 28 | 83
  Week 24: HAQ-DI score (0-3) | -19.38 [-50.0 to 3.8] | -37.50 [-58.8 to -12.5]
  Week 28: HAQ-DI score (0-3): number analyzed (Participants) | 27 | 82
  Week 28: HAQ-DI score (0-3) | -31.25 [-80.0 to 0.0] | -41.05 [-75.0 to -10.0]
  Week 32: HAQ-DI score (0-3): number analyzed (Participants) | 27 | 81
  Week 32: HAQ-DI score (0-3) | -42.86 [-75.0 to -10.0] | -41.18 [-80.0 to -12.5]
  Week 36: HAQ-DI score (0-3): number analyzed (Participants) | 27 | 81
  Week 36: HAQ-DI score (0-3) | -50.00 [-81.3 to -12.5] | -37.50 [-80.0 to -12.5]
  Week 44: HAQ-DI score (0-3): number analyzed (Participants) | 27 | 81
  Week 44: HAQ-DI score (0-3) | -57.14 [-80.0 to -25.0] | -37.50 [-80.0 to -12.5]
  Week 56: HAQ-DI score (0-3): number analyzed (Participants) | 27 | 80
  Week 56: HAQ-DI score (0-3) | -54.55 [-83.3 to -38.5] | -39.23 [-80.4 to -11.8]
  Week 24: CRP | 6.19 [-30.3 to 93.5] | -43.62 [-79.0 to 3.7]
  Week 28: CRP: number analyzed (Participants) | 28 | 84
  Week 28: CRP | -35.63 [-52.7 to -1.6] | -52.70 [-79.6 to -1.7]
  Week 32: CRP: number analyzed (Participants) | 28 | 84
  Week 32: CRP | -42.61 [-60.8 to -21.8] | -50.63 [-78.7 to -4.1]
  Week 36: CRP: number analyzed (Participants) | 28 | 85
  Week 36: CRP | -38.90 [-70.0 to -13.3] | -53.22 [-81.4 to -6.0]
  Week 44: CRP: number analyzed (Participants) | 28 | 84
  Week 44: CRP | -53.43 [-76.9 to -36.5] | -53.36 [-75.7 to -10.3]
  Week 56: CRP: number analyzed (Participants) | 28 | 84
  Week 56: CRP | -51.26 [-81.5 to -37.8] | -54.91 [-79.3 to 25.7]

12. Secondary Outcome: Change From Baseline in HAQ-DI Response at Weeks 4, 8, 12, 16, 20, and 24
Description: as for outcome 3
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
units on a scale
  Week 4 | -0.02 (0.329) | -0.17 (0.322)
  Week 8 | -0.07 (0.440) | -0.32 (0.442)
  Week 12 | -0.05 (0.450) | -0.33 (0.390)
  Week 16 | -0.05 (0.428) | -0.38 (0.397)
  Week 20 | -0.08 (0.479) | -0.41 (0.453)
  Week 24 | -0.06 (0.530) | -0.42 (0.512)

13. Secondary Outcome: Change From Baseline in HAQ-DI Score at Weeks 24, 28, 32, 36, 44, and 56
Description: Change from baseline in HAQ-DI score is a measure of the change in the physical function, where a negative change reflects an improvement and a positive change reflects worsening of physical function. HAQ-DI is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area (that is, lower scores are indicative of better functioning). The total HAQ-DI score ranges from 0-24 with lower score indicating better functioning.
Time Frame: Baseline and Weeks 24, 28, 32, 36, 44, 56
Population: Post Week 24 efficacy analysis set with observed data. Here 'n' (number analyzed) included all participants who were evaluable at specified timepoints. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
units on a scale
  Week 24 | -0.19 (0.581) | -0.46 (0.530)
  Week 28: number analyzed (Participants) | 28 | 85
  Week 28 | -0.40 (0.646) | -0.51 (0.571)
  Week 32: number analyzed (Participants) | 28 | 84
  Week 32 | -0.50 (0.624) | -0.56 (0.595)
  Week 36: number analyzed (Participants) | 28 | 84
  Week 36 | -0.59 (0.650) | -0.53 (0.618)
  Week 44: number analyzed (Participants) | 28 | 84
  Week 44 | -0.63 (0.612) | -0.54 (0.598)
  Week 56: number analyzed (Participants) | 28 | 83
  Week 56 | -0.67 (0.558) | -0.55 (0.621)

14. Secondary Outcome: Percentage of Participants Who Achieved a HAQ-DI Response With Greater Than or Equal to (>=) 0.3 Improvement From Baseline in HAQ-DI Score at Weeks 4, 8, 12, 16, 20, and 24
Description: HAQ-DI response was defined as >= 0.3 improvement from baseline in HAQ-DI score. HAQ-DI is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0 indicating no difficulty, to 3 indicating inability to perform a task in that area (that is, lower scores are indicative of better functioning). The total HAQ-DI score ranges from 0-24 with lower score indicating better functioning.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
percentage of participants
  Week 4 | 12.2 | 29.0
  Week 8 | 26.5 | 43.0
  Week 12 | 22.4 | 47.0
  Week 16 | 20.4 | 50.0
  Week 20 | 22.4 | 48.0
  Week 24 | 28.6 | 51.0

15. Secondary Outcome: Percentage of Participants Who Achieved an HAQ-DI Response With >= -0.3 Improvement From Baseline in HAQ-DI Score at Weeks 24, 28, 32, 36, 44, and 56
Description: HAQ-DI response was defined as >= 0.3 improvement from baseline in HAQ-DI score. HAQ-DI is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0 indicating no difficulty, to 3 indicating inability to perform a task in that area (that is, lower scores are indicative of better functioning). The total HAQ-DI score ranges from 0-24 with lower score indicating better functioning. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Time Frame: Weeks 24, 28, 32, 36, 44, 56
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
percentage of participants
  Week 24 | 44.8 | 55.8
  Week 28: number analyzed (Participants) | 28 | 85
  Week 28 | 53.6 | 60.0
  Week 32: number analyzed (Participants) | 28 | 84
  Week 32 | 57.1 | 56.0
  Week 36: number analyzed (Participants) | 28 | 84
  Week 36 | 64.3 | 59.5
  Week 44: number analyzed (Participants) | 28 | 84
  Week 44 | 71.4 | 61.9
  Week 56: number analyzed (Participants) | 28 | 83
  Week 56 | 75.0 | 59.0

16. Secondary Outcome: Percent Change From Baseline in Dactylitis Scores at Weeks 4, 8, 16, and 24
Description: as for outcome 7
Time Frame: Baseline and Weeks 4, 8, 16, 24
Population: FAS (up to week 24) and who had dactylitis at baseline. Data after EE to ustekinumab or missing data were imputed using LOCF. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 23 | 58
percent change
  Week 4 | -33.33 [-50.0 to 0.0] | -32.46 [-100.0 to 0.0]
  Week 8 | -50.00 [-75.00 to 0.0] | -75.00 [-100.0 to -10.0]
  Week 16 | -50.00 [-80.0 to 0.0] | -100.00 [-100.0 to -33.3]
  Week 24 | -33.33 [-66.7 to 0.0] | -100.00 [-100.00 to -50.0]

17. Secondary Outcome: Percent Change From Baseline in Dactylitis Scores at Weeks 24, 28, 32, 44, 56
Description: Dactylitis was characterized by swelling of the entire finger or toe. The severity of dactylitis is scored on a scale of 0-3, where 0, 1, 2, 3 indicates none, mild, moderate, severe, respectively in each digit of the hands and feet. The range of total dactylitis scores for a participant is 0-60. Higher score indicates more severe dactylitis. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Time Frame: Baseline and Weeks 24, 28, 32, 44, 56
Population: Post Week 24 efficacy analysis set with observed data and who had dactylitis at baseline. Here 'n' (number analyzed) included all participants who were evaluable at specified timepoints. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 16 | 50
percent change
  Week 24 | -45.00 [-70.8 to 0.0] | -100.00 [-100.0 to -80.0]
  Week 28: number analyzed (Participants) | 16 | 49
  Week 28 | -70.83 [-100.0 to -22.5] | -100.00 [-100.00 to -66.7]
  Week 32: number analyzed (Participants) | 16 | 49
  Week 32 | -100.00 [-100.00 to -79.2] | -100.00 [-100.00 to -70.0]
  Week 44: number analyzed (Participants) | 16 | 49
  Week 44 | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]
  Week 56: number analyzed (Participants) | 16 | 48
  Week 56 | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -95.0]

18. Secondary Outcome: Percentage of Participants With Dactylitis at Weeks 4, 8, 16, and 24
Description: Dactylitis is characterized by swelling of the entire finger or toe. The severity of dactylitis is scored on a scale of 0-3, where 0, 1, 2, 3 indicates none, mild, moderate, severe, respectively in each digit of the hands and feet. The range of total dactylitis scores for a participant is 0-60. Participants with dactylitis had dactylitis score >0. Higher score indicates more severe dactylitis.
Time Frame: Weeks 4, 8, 16, and 24
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 23 | 58
percentage of participants
  Week 4 | 91.3 | 72.4
  Week 8 | 69.6 | 56.9
  Week 16 | 78.3 | 48.3
  Week 24 | 82.6 | 44.8

19. Secondary Outcome: Percentage of Participants With Dactylitis at Weeks 24, 28, 32, 44, and 56
Description: Dactylitis was characterized by swelling of the entire finger or toe. The severity of dactylitis is scored on a scale of 0-3, where 0, 1, 2, 3 indicates none, mild, moderate, severe, respectively in each digit of the hands and feet. The range of total dactylitis scores for a participant is 0-60. Higher score indicates greater degree of tenderness.
Time Frame: Weeks 24, 28, 32, 44, and 56
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 16 | 50
percentage of participants
  Week 24 | 81.3 | 40.0
  Week 28: number analyzed (Participants) | 16 | 49
  Week 28 | 62.5 | 38.8
  Week 32: number analyzed (Participants) | 16 | 49
  Week 32 | 31.3 | 36.7
  Week 44: number analyzed (Participants) | 16 | 49
  Week 44 | 12.5 | 20.4
  Week 56: number analyzed (Participants) | 16 | 48
  Week 56 | 6.3 | 25.0

20. Secondary Outcome: Percent Change From Baseline in LEI Scores at Week 4, 8, 16, and 24
Description: as for outcome 6
Time Frame: Baseline and Weeks 4, 8, 16, 24
Population: FAS (up to Week 24) and who had enthesitis at baseline. Data after EE to ustekinumab or missing data are imputed using LOCF. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 31 | 76
percent change
  Week 4 | 0.00 [-50.0 to 0.0] | -18.33 [-79.2 to 0.0]
  Week 8 | 0.00 [-60.0 to 0.0] | -58.33 [-100.0 to 0.0]
  Week 16 | 0.00 [-50.0 to 0.00] | -50.04 [-100.0 to 0.00]
  Week 24 | -33.33 [-100.00 to 0.0] | -100.00 [-100.00 to 0.0]

21. Secondary Outcome: Percent Change From Baseline in LEI Scores at Weeks 24, 28, 32, 44, and 56
Description: Enthesitis will be assessed using the Leeds Enthesitis Index (LEI). The LEI was developed to assess enthesitis in participants with PsA, and evaluates the presence (score of 1) or absence of pain (score of 0) by applying local pressure to Lateral elbow epicondyle, left and right, Medial femoral condyle, left and right, and Achilles tendon insertion, left and right. LEI scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness).
Time Frame: Baseline and Weeks 24, 28, 32, 44, 56
Population: Post Week 24 efficacy analysis set with observed data and who had enthesitis at baseline. Here 'n' (number analyzed) included all participants who were evaluable at specified timepoints. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 18 | 67
percent change
  Week 24 | -50.00 [-100.0 to 0.0] | -100.00 [-100.0 to -50.0]
  Week 28: number analyzed (Participants) | 17 | 67
  Week 28 | -60.00 [-100.0 to -40.0] | -100.00 [-100.0 to -50.0]
  Week 32: number analyzed (Participants) | 17 | 66
  Week 32 | -100.00 [-100.0 to -60.0] | -100.00 [-100.0 to -66.7]
  Week 44: number analyzed (Participants) | 17 | 66
  Week 44 | -100.00 [-100.0 to -60.0] | -100.00 [-100.0 to -50.0]
  Week 56: number analyzed (Participants) | 16 | 65
  Week 56 | -100.00 [-100.0 to -35.0] | -100.00 [-100.0 to -50.0]

22. Secondary Outcome: Percentage of Participants With Enthesitis Based on LEI Score at Weeks 4, 8, 16, and 24 in Participants With Enthesitis at Baseline
Description: Enthesitis was assessed using the Leeds Enthesitis Index (LEI). The LEI was developed to assess enthesitis in participants with PsA, and evaluates the presence (score of 1) or absence of pain (score of 0) by applying local pressure to Lateral elbow epicondyle, left and right, Medial femoral condyle, left and right, and Achilles tendon insertion, left and right. Participants with enthesitis had LEI score >0. LEI scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness).
Time Frame: Weeks 4, 8, 16, and 24
Population: FAS (up to Week 24) and who had enthesitis at baseline. Data after EE to ustekinumab or missing data were imputed using LOCF. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Number; unit: percentage of Participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 31 | 76
percentage of Participants
  Week 4 | 87.1 | 76.3
  Week 8 | 87.1 | 59.2
  Week 16 | 83.9 | 53.9
  Week 24 | 71.0 | 43.4

23. Secondary Outcome: Percentage of Participants With Enthesitis Based on LEI at Weeks 24, 28, 32, 44, and 56 in Participants With Enthesitis at Baseline
Description: Enthesitis will be assessed using the Leeds Enthesitis Index (LEI). The LEI was developed to assess enthesitis in participants with PsA, and evaluates the presence (score of 1) or absence of pain (score of 0) by applying local pressure to Lateral elbow epicondyle, left and right, Medial femoral condyle, left and right, and Achilles tendon insertion, left and right. Participants with enthesitis had LEI score >0. LEI scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness).
Time Frame: Weeks 24, 28, 32, 44, and 56
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 18 | 67
percentage of participants
  Week 24 | 66.7 | 38.8
  Week 28: number analyzed (Participants) | 17 | 67
  Week 28 | 64.7 | 44.8
  Week 32: number analyzed (Participants) | 17 | 66
  Week 32 | 35.3 | 31.8
  Week 44: number analyzed (Participants) | 17 | 66
  Week 44 | 47.1 | 37.9
  Week 56: number analyzed (Participants) | 16 | 65
  Week 56 | 37.5 | 29.2

24. Secondary Outcome: Change From Baseline in Psoriatic ArthritiS Disease Activity Score (PASDAS) Score at Weeks 16 and 24
Description: Change from baseline in PASDAS score measures the change in disease activity where a negative value indicates an improvement and a positive value indicates worsening of PsA disease activity. PASDAS is a PsA disease activity score that assesses 4 domains (joints, entheses, dactylitis and quality of life) of PsA. PASDAS is a derived score combining Patient's Global Assessment of Disease Activity (arthritis and psoriasis, on a 100-unit VAS), Physician's Global Assessment of Disease Activity (on a 100-unit VAS), swollen joint count (66 joints), tender joint count (68 joints), CRP (mg/L), enthesitis based on LEI (scaled to a 0-6 range), dactylitis count (scoring each digit from 0-3 and recoding to 0-1, where any score > 0 equaled 1), and the PCS score of the SF-36 health survey. The total score range is 0-10 and the cutoffs for disease activity were 3.2 (low) to 5.4 (high). Negative changes from baseline indicate improvement of overall disease activity.
Time Frame: Baseline and Weeks 16, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
units on a scale
  Week 16 | -0.45 (1.099) | -2.24 (1.458)
  Week 24 | -0.49 (1.333) | -2.50 (1.587)

25. Secondary Outcome: Change From Baseline in PASDAS Score at Weeks 24 and 44
Description: as for outcome 24
Time Frame: Baseline and Weeks 24, 44
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
units on a scale
  Week 24: number analyzed (Participants) | 28 | 86
  Week 24 | -1.05 (1.440) | -2.80 (1.454)
  Week 44: number analyzed (Participants) | 28 | 83
  Week 44 | -3.17 (1.524) | -3.15 (1.570)

26. Secondary Outcome: Change From Baseline in GRAppa Composite scorE (GRACE) Index Score at Weeks 16 and 24
Description: Change from baseline in GRACE index score measures the change in disease activity, where a negative change indicates an improvement and a positive change indicates a worsening of PsA disease activity. GRACE index was converted from Arithmetic Mean of the Desirability Function (AMDF). AMDF is calculated by transforming all variables using predefined algorithms and expressing the total score as a mean with a score range of 0 - 1, where 1 indicates a better state than 0. GRACE Index = (1 - AMDF)*10, where GRACE index has a range of 0-10, with higher scores indicate more active disease. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Time Frame: Baseline and Weeks 16, 24
Population: FAS (up to Week 24). Data after EE to ustekinumab and missing data were imputed using LOCF. Here 'N' (number of participants analyzed) included all participants who were evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 48 | 98
units on a scale
  Week 16 | -0.29 (1.174) | -2.49 (1.614)
  Week 24 | -0.35 (1.394) | -2.73 (1.756)

27. Secondary Outcome: Change From Baseline in GRACE Index Score at Weeks 24 and 44
Description: Change from baseline in GRACE index score measures the change in disease activity, where a negative change indicates an improvement and a positive change indicates a worsening of PsA disease activity. GRACE index was converted from Arithmetic Mean of the Desirability Function (AMDF). AMDF is calculated by transforming all variables using predefined algorithms and expressing the total score as a mean with a score range of 0 - 1, where 1 indicates a better state than 0. GRACE Index = (1 - AMDF)*10, where GRACE index has a range of 0-10, with higher scores indicate more active disease.
Time Frame: Baseline and Weeks 24, 44
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
units on a scale
  Week 24: number analyzed (Participants) | 27 | 85
  Week 24 | -0.91 (1.498) | -2.96 (1.717)
  Week 44: number analyzed (Participants) | 27 | 82
  Week 44 | -3.21 (1.698) | -3.26 (1.856)

28. Secondary Outcome: Change From Baseline in Modified Composite Psoriatic Disease Activity Index (mCPDAI) Score at Weeks 16 and 24
Description: The mCPDAI assessed 4 domains (joints, skin, entheses, and dactylitis). The mCPDAI scores were calculated using the following assessments: joints (66 swollen and 68 tender joint counts), HAQ-DI score, PASI, dactylitis, and enthesitis. Within each domain a score (range 0-3) was assigned, where 0= Not involved, 1= Mild, 2= Moderate and 3= Severe. The scores for each domain were then added together to give a final score range of 0 to 12. A higher score indicates more active disease activity. Negative changes from baseline indicate improvement of PsA disease activity.
Time Frame: Baseline and Weeks 16, 24
Population: FAS (up to Week 24). Data after EE to ustekinumab and missing data were imputed using LOCF. Here 'N' (number of participants analyzed) included all participants who were evaluable for this endpoint. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 48 | 98
units on a scale
  Week 16 | -0.5 (1.88) | -3.1 (2.48)
  Week 24 | -0.8 (2.16) | -3.9 (2.72)

29. Secondary Outcome: Change From Baseline in mCPDAI Index Score at Weeks 24 and 44
Description: as for outcome 28
Time Frame: Baseline and Weeks 24, 44
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo to Guselkumab (CO) at Week 24: Participants who were randomized to receive placebo matched to guselkumab at Weeks 0, 4, 12 and 20 received guselkumab 100 mg subcutaneous injection at Weeks 24, 28, 36 and 44.
Arm/Group | Placebo to Guselkumab (CO) at Week 24 | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
units on a scale
  Week 24: number analyzed (Participants) | 27 | 85
  Week 24 | -1.4 (2.27) | -4.3 (2.69)
  Week 44: number analyzed (Participants) | 27 | 82
  Week 44 | -4.2 (2.88) | -4.8 (2.55)

30. Secondary Outcome: Change From Baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) Score at Weeks 4, 8, 12, 16, 20 and 24
Description: Change from baseline in DAPSA measures the change in disease activity, where a negative change indicates an improvement and a positive change indicates worsening of disease activity. DAPSA score is a the sum of swollen joint count (66 joints), tender joint count (68 joints), CRP (mg/dL), Patient's Assessment of Pain (on a 10-unit VAS;0=no pain, 10=worst possible pain), and Patient's Global Assessment of Disease Activity (arthritis, on a 10-unit VAS; 0 to 100 centimeter [cm] VAS, 0=excellent and 10=poor). Cut-off values for disease activity: 0-4 remission; 5-14 low; 15-28 moderate; >28 high.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24
Population: FAS (up to Week 24). Data after early escape (EE) to ustekinumab and missing data were imputed using LOCF. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Guselkumab: Participants were randomized to receive guselkumab 100 mg subcutaneous injections at Weeks 0, 4, 12, 20, 28, 36 and 44, and matched placebo at Week 24.
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
units on a scale
  Week 4 | -5.62 (13.030) | -10.03 (11.207)
  Week 8 | -8.25 (15.158) | -16.65 (15.948)
  Week 12 | -6.84 (16.334) | -18.84 (16.266)
  Week 16 | -4.98 (16.045) | -21.26 (17.811)
  Week 20 | -4.70 (17.408) | -22.56 (19.918)
  Week 24 | -4.97 (20.114) | -23.08 (20.206)

31. Secondary Outcome: Change From Baseline in DAPSA Index Score at Weeks 24, 28, 32, 36, 44, and 56
Description: Change from baseline in DAPSA measures the change in disease activity, where a negative change indicates an improvement and a positive change indicates worsening of disease activity. DAPSA score is a the sum of swollen joint count (66 joints), tender joint count (68 joints), CRP (mg/dL), Patient's Assessment of Pain (on a 10-unit VAS;0=no pain, 10=worst possible pain), and Patient's Global Assessment of Disease Activity (arthritis, on a 10-unit VAS; 0 to 10cm VAS, 0=excellent and 10=poor). Cut-off values for disease activity: 0-4 remission; 5-14 low; 15-28 moderate; >28 high.
Time Frame: Baseline and Weeks 24, 28, 32, 36, 44, 56
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
units on a scale
  Week 24 | -12.99 (22.328) | -26.93 (18.238)
  Week 28: number analyzed (Participants) | 28 | 85
  Week 28 | -20.85 (21.434) | -29.71 (18.911)
  Week 32: number analyzed (Participants) | 28 | 84
  Week 32 | -26.12 (21.309) | -30.59 (19.720)
  Week 36: number analyzed (Participants) | 28 | 85
  Week 36 | -27.37 (22.480) | -30.43 (18.114)
  Week 44: number analyzed (Participants) | 28 | 84
  Week 44 | -29.54 (20.785) | -30.55 (18.188)
  Week 56: number analyzed (Participants) | 28 | 84
  Week 56 | -31.98 (20.359) | -32.02 (18.328)

32. Secondary Outcome: Percentage of Participants Who Achieved Minimal Disease Activity (MDA) at Weeks 16 and 24
Description: MDA defines a satisfactory state of disease activity that includes 5 domains of PsA (joint symptoms, skin psoriasis, patient's perspective of pain and disease activity on arthritis and psoriasis, physical function and enthesitis). Participants were classified as achieving MDA if they fulfilled 5 of 7 outcome measures: tender joint count <=1; swollen joint count <=1; PASI <=1; patient pain VAS score of <=15 mm; patient global disease activity on arthritis and psoriasis; VAS score of <=20 mm; Health Assessment Questionnaire score <=0.5; and tender entheseal points <=1.
Time Frame: Weeks 16 and 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
percentage of participants
  Week 16 | 0 | 18.0
  Week 24 | 2.0 | 23.0

33. Secondary Outcome: Percentage of Participants Who Achieved MDA at Weeks 24 and 44
Description: as for outcome 32
Time Frame: Weeks 24 and 44
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
percentage of participants
  Week 24 | 3.4 | 26.7
  Week 44: number analyzed (Participants) | 28 | 84
  Week 44 | 28.6 | 34.5

34. Secondary Outcome: Change From Baseline in the Physical and Mental Component Summary (PCS and MCS) Scores of 36- Item Short Form Health Assessment Questionnaire (SF-36) at Weeks 16 and 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The PCS and MCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms as presented in this outcome measure. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline and Weeks 16, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
units on a scale
  Week 16: PCS | -0.44 (5.025) | 5.86 (7.315)
  Week 24: PCS | 0.46 (6.513) | 6.59 (7.465)
  Week 16: MCS | 1.14 (7.075) | 4.80 (8.952)
  Week 24: MCS | 0.42 (6.737) | 4.95 (9.064)

35. Secondary Outcome: Change From Baseline in the PCS Scores of SF-36 at Weeks 24 and 44
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The PCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms as presented in this outcome measure. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline and Weeks 24, 44
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
units on a scale
  Week 24: PCS: number analyzed (Participants) | 28 | 86
  Week 24: PCS | 2.13 (7.365) | 7.40 (7.448)
  Week 44: PCS: number analyzed (Participants) | 28 | 84
  Week 44: PCS | 8.02 (8.647) | 8.34 (8.783)

36. Secondary Outcome: Change From Baseline in the MCS Scores of SF-36 at Weeks 24 and 44
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The MCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms as presented in this outcome measure. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline and Weeks 24, 44
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
units on a scale
  Week 24: MCS: number analyzed (Participants) | 28 | 86
  Week 24: MCS | 0.51 (6.770) | 5.45 (9.081)
  Week 44: MCS: number analyzed (Participants) | 28 | 84
  Week 44: MCS | 5.53 (9.013) | 4.56 (9.548)

37. Secondary Outcome: Change From Baseline in Norm-based SF-36 Scales at Week 16 and 24
Description: SF-36 evaluates 8 individual subscales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health). Each 8 scales scored from 0 to 100 with higher scores= better health. The scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. Higher scores indicate better health. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline and Weeks 16, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
T-score
  Week 16: Physical functioning | -0.31 (6.657) | 6.30 (7.255)
  Week 24: Physical functioning | -0.04 (8.227) | 6.93 (8.009)
  Week 16: Role-physical | -0.23 (5.674) | 4.22 (7.146)
  Week 24: Role-physical | -0.09 (6.813) | 4.69 (7.961)
  Week 16: Bodily pain | 0.21 (5.675) | 6.56 (7.832)
  Week 24: Bodily pain | 0.81 (6.445) | 7.56 (8.288)
  Week 16: General health | 0.74 (5.857) | 6.19 (7.964)
  Week 24: General health | 1.49 (7.274) | 6.48 (7.676)
  Week 16: Vitality | 0.73 (7.779) | 5.85 (8.138)
  Week 24: Vitality | 1.46 (7.254) | 6.39 (8.861)
  Week 16: Social functioning | -0.82 (8.272) | 5.87 (9.346)
  Week 24: Social functioning | -0.82 (7.613) | 6.22 (10.426)
  Week 16: Role-emotional | 1.14 (8.774) | 4.77 (9.643)
  Week 24: Role-emotional | 0.64 (8.754) | 4.67 (9.393)
  Week 16: Mental health | 1.28 (7.007) | 5.10 (8.683)
  Week 24: Mental health | 0.21 (7.020) | 5.68 (8.877)

38. Secondary Outcome: Change From Baseline in Norm-based SF-36 Scale at Week 24 and 44
Description: as for outcome 37
Time Frame: Baseline and Weeks 24, 44
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
T-score
  Week 24: Physical functioning: number analyzed (Participants) | 28 | 86
  Week 24: Physical functioning | 1.09 (8.953) | 7.54 (8.228)
  Week 44: Physical functioning: number analyzed (Participants) | 28 | 84
  Week 44: Physical functioning | 8.41 (9.969) | 8.50 (8.633)
  Week 24: Role-physical: number analyzed (Participants) | 28 | 86
  Week 24: Role-physical | 1.92 (7.119) | 5.74 (7.480)
  Week 44: Role-physical: number analyzed (Participants) | 28 | 84
  Week 44: Role-physical | 6.82 (9.198) | 6.66 (7.664)
  Week 24: Bodily pain: number analyzed (Participants) | 28 | 86
  Week 24: Bodily pain | 2.88 (6.856) | 8.39 (8.332)
  Week 44: Bodily pain: number analyzed (Participants) | 28 | 84
  Week 44: Bodily pain | 9.42 (8.914) | 8.95 (9.952)
  Week 24: General health: number analyzed (Participants) | 28 | 86
  Week 24: General health | 1.94 (8.185) | 7.05 (7.657)
  Week 44: General health: number analyzed (Participants) | 28 | 84
  Week 44: General health | 6.25 (8.998) | 6.74 (8.496)
  Week 24: Vitality: number analyzed (Participants) | 28 | 86
  Week 24: Vitality | 1.49 (7.387) | 7.39 (8.727)
  Week 44: Vitality: number analyzed (Participants) | 28 | 84
  Week 44: Vitality | 7.53 (10.802) | 7.11 (9.891)
  Week 24: Social functioning: number analyzed (Participants) | 28 | 86
  Week 24: Social functioning | -0.18 (7.776) | 6.41 (10.919)
  Week 44: Social functioning: number analyzed (Participants) | 28 | 84
  Week 44: Social functioning | 6.09 (10.151) | 5.73 (10.357)
  Week 24: Role-emotional: number analyzed (Participants) | 28 | 86
  Week 24: Role-emotional | 2.11 (7.891) | 5.30 (9.013)
  Week 44: Role-emotional: number analyzed (Participants) | 28 | 84
  Week 44: Role-emotional | 5.47 (9.160) | 5.68 (9.635)
  Week 24: Mental health: number analyzed (Participants) | 28 | 86
  Week 24: Mental health | 0.19 (7.465) | 6.30 (8.994)
  Week 44: Mental health: number analyzed (Participants) | 28 | 84
  Week 44: Mental health | 7.29 (9.952) | 5.42 (8.978)

39. Secondary Outcome: Change From Baseline in Routine Assessment of Patient Index Data 3 (RAPID3) Score at Weeks 16 and 24
Description: RAPID3 is a multi-dimensional health assessment questionnaire that was designed for use in routine clinical care. Three core data set for function, pain, and patient global estimate of disease activity were recorded. Each was scored 0-10 and the score ranges from 0 to 30 with higher scores indicating worse condition. A negative change from baseline indicates improvement in condition.
Time Frame: Baseline and Weeks 16, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 49 | 100
units on a scale
  Week 16 | -0.19 (4.405) | -5.41 (5.307)
  Week 24 | -0.57 (5.123) | -5.81 (5.968)

40. Secondary Outcome: Change From Baseline in RAPID3 Score at Weeks 24 and 44
Description: as for outcome 39
Time Frame: Baseline and Weeks 24, 44
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab (CO) at Week 24 | Guselkumab
Number analyzed (Participants) | 29 | 86
units on a scale
  Week 24: number analyzed (Participants) | 28 | 86
  Week 24 | -2.28 (5.244) | -6.36 (6.205)
  Week 44: number analyzed (Participants) | 28 | 84
  Week 44 | -7.60 (6.588) | -7.48 (6.310)

41. Secondary Outcome: Percentage of Participants Who Achieved a PASI 50, PASI 75, PASI 90 and PASI 100 Response at Weeks 16 and 24
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. PASI 50, 75, 90, and 100 responses were defined as at least a 50%, 75%, 90%, and 100% reduction in PASI relative to Baseline respectively. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Time Frame: Weeks 16 and 24
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 48 | 98
percentage of participants
  Week 16: PASI 50 responders | 27.1 | 81.6
  Week 16: PASI 75 responders | 8.3 | 71.4
  Week 16: PASI 90 responders | 6.3 | 53.1
  Week 16: PASI 100 responders | 6.3 | 31.6
  Week 24: PASI 50 responders | 29.2 | 86.7
  Week 24: PASI 75 responders | 12.5 | 78.6
  Week 24: PASI 90 responders | 6.3 | 66.3
  Week 24: PASI 100 responders | 6.3 | 39.8

42. Secondary Outcome: Percentage of Participants Who Achieved a PASI 50, PASI 75, PASI 90 and PASI 100 Response at Weeks 24, 28, 32, 44, and 56
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. PASI 50, 75, 90, and 100 responses were defined as at least a 50%, 75%, 90%, and 100% reduction in PASI relative to Baseline respectively.
Time Frame: Weeks 24, 28, 32, 44, and 56
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
percentage of participants
  Week 24: PASI 50 responders | 37.9 | 89.5
  Week 24: PASI 75 responders | 20.7 | 82.6
  Week 24: PASI 90 responders | 10.3 | 70.9
  Week 24: PASI 100 responders | 10.3 | 44.2
  Week 28: PASI 50 responders: number analyzed (Participants) | 28 | 84
  Week 28: PASI 50 responders | 60.7 | 95.2
  Week 28: PASI 75 responders: number analyzed (Participants) | 28 | 84
  Week 28: PASI 75 responders | 35.7 | 84.5
  Week 28: PASI 90 responders: number analyzed (Participants) | 28 | 84
  Week 28: PASI 90 responders | 25.0 | 72.6
  Week 28: PASI 100 responders: number analyzed (Participants) | 28 | 84
  Week 28: PASI 100 responders | 17.9 | 53.6
  Week 32: PASI 50 responders: number analyzed (Participants) | 28 | 83
  Week 32: PASI 50 responders | 78.6 | 92.8
  Week 32: PASI 75 responders: number analyzed (Participants) | 28 | 83
  Week 32: PASI 75 responders | 67.9 | 86.7
  Week 32: PASI 90 responders: number analyzed (Participants) | 28 | 83
  Week 32: PASI 90 responders | 50.0 | 80.7
  Week 32: PASI 100 responders: number analyzed (Participants) | 28 | 83
  Week 32: PASI 100 responders | 35.7 | 62.7
  Week 44: PASI 50 responders: number analyzed (Participants) | 28 | 83
  Week 44: PASI 50 responders | 89.3 | 94.0
  Week 44: PASI 75 responders: number analyzed (Participants) | 28 | 83
  Week 44: PASI 75 responders | 82.1 | 90.4
  Week 44: PASI 90 responders: number analyzed (Participants) | 28 | 83
  Week 44: PASI 90 responders | 75.0 | 81.9
  Week 44: PASI 100 responders: number analyzed (Participants) | 28 | 83
  Week 44: PASI 100 responders | 67.9 | 63.9
  Week 56: PASI 50 responders: number analyzed (Participants) | 27 | 82
  Week 56: PASI 50 responders | 96.3 | 92.7
  Week 56: PASI 75 responders: number analyzed (Participants) | 27 | 82
  Week 56: PASI 75 responders | 81.5 | 85.4
  Week 56: PASI 90 responders: number analyzed (Participants) | 27 | 82
  Week 56: PASI 90 responders | 74.1 | 78.0
  Week 56: PASI 100 responders: number analyzed (Participants) | 27 | 82
  Week 56: PASI 100 responders | 55.6 | 57.3

43. Secondary Outcome: Percent Change From Baseline in PASI Score at Weeks 4, 8, 16, and 24
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A negative percent change from baseline indicates the percent improvement from baseline in the severity of psoriatic lesions. As planned, results data was analyzed and reported for the specified arms for this outcome measure.
Time Frame: Baseline and Weeks 4, 8, 16, 24
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 48 | 98
percent change
  Week 4 | 0.00 [-16.0 to 17.0] | -41.49 [-64.7 to -12.2]
  Week 8 | 1.58 [-20.2 to 24.9] | -66.67 [-93.6 to -41.9]
  Week 16 | -1.10 [-50.0 to 35.9] | -90.55 [-100.0 to -65.6]
  Week 24 | -7.89 [-54.2 to 34.0] | -96.21 [-100.0 to -82.6]

44. Secondary Outcome: Percent Change From Baseline in PASI Score at Weeks 24, 28, 32, 44, and 56
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A negative percent change from baseline indicates the percent improvement from baseline in the severity of psoriatic lesions.
Time Frame: Baseline and Weeks 24, 28, 32, 44, 56
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 24 to Week 52)
Number analyzed (Participants) | 29 | 86
percent change
  Week 24: number analyzed (Participants) | 28 | 85
  Week 24 | -34.26 [-72.9 to 26.9] | -97.85 [-100.0 to -87.2]
  Week 28: number analyzed (Participants) | 27 | 83
  Week 28 | -57.69 [-94.3 to -39.4] | -100.00 [-100.0 to -88.2]
  Week 32: number analyzed (Participants) | 27 | 82
  Week 32 | -90.61 [-100.0 to -62.5] | -100.00 [-100.0 to -94.0]
  Week 44: number analyzed (Participants) | 27 | 82
  Week 44 | -100.00 [-100.0 to -91.0] | -100.00 [-100.0 to -95.4]
  Week 56: number analyzed (Participants) | 26 | 81
  Week 56 | -100.00 [-100.0 to -91.0] | -100.00 [-100.0 to -91.4]

ADVERSE EVENTS:
Time Frame: Up to Week 56
Description: The safety analysis set included all participants who received at least 1 (partial or complete) dose of study agent and were analyzed based on the actual treatment received.
Groups:
- Placebo (Week 0 to Week 24): Participants received placebo matched to guselkumab subcutaneous injections at Weeks 0, 4, 12 and 20. Data through Week 24 prior to receiving guselkumab or through Week 16 prior to receiving ustekinumab (for participants who early escaped at week 16) were included.
- Placebo to Guselkumab (Week 24 to Week 56): Participants who received placebo matched to guselkumab subcutaneous injections at Weeks 0, 4, 12 and 20 received guselkumab 100 mg subcutaneous injections at Week 24, 28, 36 and 44. Data from the first administration of guselkumab (Week 24) through Week 56 (final follow-up) were included.
- Guselkumab (Week 0 to Week 56): Participants received guselkumab 100 mg subcutaneous injections at Weeks 0, 4, 12, 20, 28, 36 and 44, and matched placebo at Week 24. Data from Week 0 through Week 56 (final follow-up) or through Week 16 prior to receiving ustekinumab (for participants who early escaped at week 16) were included.
- Placebo to Ustekinumab (EE: Week 16 to Week 56): Participants who received placebo matched to guselkumab subcutaneous injections at Weeks 0, 4, 12 and were qualified to early escape (EE) at Week 16 received open-label ustekinumab subcutaneous injections at Weeks 16, 20, 32 and 44 at the approved dosage for PsA in the particular country of the study. Data from the first administration of ustekinumab (Week 16) through Week 56 (final follow-up) were included.
- Guselkumab to Ustekinumab (EE:Week 16 to Week 56): Participants who received guselkumab subcutaneous injections at Weeks 0, 4, 12 and were qualified to early escape (EE) at Week 16 received open-label ustekinumab subcutaneous injections at Weeks 16, 20, 32 and 44 at the approved dosage for PsA in the particular country of the study. Data from the first administration of ustekinumab (Week 16) through Week 56 (final follow-up) were included.
Arm/Group | Placebo (Week 0 to Week 24) | Placebo to Guselkumab (Week 24 to Week 56) | Guselkumab (Week 0 to Week 56) | Placebo to Ustekinumab (EE: Week 16 to Week 56) | Guselkumab to Ustekinumab (EE:Week 16 to Week 56)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/29 | 0/100 | 0/17 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/29 | 6/100 | 0/17 | 0/10
Other Adverse Events (participants affected / at risk) | 7/49 | 3/29 | 24/100 | 8/17 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0 to Week 24) (N=49) | Placebo to Guselkumab (Week 24 to Week 56) (N=29) | Guselkumab (Week 0 to Week 56) (N=100) | Placebo to Ustekinumab (EE: Week 16 to Week 56) (N=17) | Guselkumab to Ustekinumab (EE:Week 16 to Week 56) (N=10)
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pupils Unequal (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ulcerative Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0 to Week 24) (N=49) | Placebo to Guselkumab (Week 24 to Week 56) (N=29) | Guselkumab (Week 0 to Week 56) (N=100) | Placebo to Ustekinumab (EE: Week 16 to Week 56) (N=17) | Guselkumab to Ustekinumab (EE:Week 16 to Week 56) (N=10)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 5 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 0 | 10 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 2 | 4 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 2 | 3 | 0 | 1
Weight Increased (Investigations) | 1 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Depressive Symptom (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.